CLINICAL TRIAL: NCT00464438
Title: A Study to Evaluate the Safety and Efficacy of Gatifloxacin for the Treatment of Bacterial Conjunctivitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Therapeutic Area Head, Allergan, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 198782-003
Record Dates: First submitted 2007-04-19; First posted 2007-04-23 (Estimated); Results first posted 2011-09-21 (Estimated); Last update posted 2011-09-21 (Estimated); Status verified 2011-08

CONDITIONS: Bacterial Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Bacterial | interventions — Gatifloxacin; Moxifloxacin; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: gatifloxacin
- 2 (Active Comparator)
  Interventions: Drug: gatifloxacin; Drug: moxifloxacin 0.5% eye drops

INTERVENTIONS:
Drug: gatifloxacin — Day 1-6 = 1 drop of study medication three times a day
  Other Names: Zymar®
Drug: moxifloxacin 0.5% eye drops — Day 1-6 = 1 drop of study medication three times a day
  Other Names: Vigamox®
  Arms: 2

SUMMARY:
This is a 7 day study to evaluate the safety and efficacy of topical gatifloxacin ophthalmic solution for the treatment of bacterial conjunctivitis in subjects from birth to 31 days of age

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with bacterial conjunctivitis

Exclusion Criteria:

* chemical or foreign body trauma to either eye
* infection in either eye (besides bacterial conjunctivitis)
* white spots in the cornea or ulcers in either eye
* clinical diagnosis of chlamydia or gonorrhea in either eye

Max Age: 31 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 171 (Actual)
Dates: Start 2007-06; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (2):
- Sacramento, California, United States
- Whitby, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gatifloxacin 0.3% | Moxifloxacin 0.5%
Started | 85 | 86
Completed | 83 | 80
Not Completed | 2 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gatifloxacin 0.3% | Moxifloxacin 0.5% | Total
Number analyzed (Participants) | 85 | 86 | 171
Age Continuous [Mean (Standard Deviation); unit: days] | 15.2 (6.59) | 15.2 (6.05) | 15.2 (6.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 22 | 59
  Male | 48 | 64 | 112

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Clearing (Clinical Success) of Conjunctival Erythema and Conjunctival Discharge at Day 7
Description: Percentage of patients that achieved clinical success, defined as a score of 0 for both conjunctival erythema and conjunctival discharge at Day 7. Conjunctival erythema and conjunctival discharge were each assessed on a 4-point severity grade scale (0=none, +1=mild, +2=moderate, +3=severe).
Time Frame: Day 7
Population: Modified Intent to Treat; defined as all randomized patients who were "culture positive" at baseline meaning the culture of the eye grew bacteria.
Measure: Number; unit: Percentage of Patients
Arm/Group | Gatifloxacin 0.3% | Moxifloxacin 0.5%
Number analyzed (Participants) | 56 | 64
Percentage of Patients | 78.6 | 84.4

2. Secondary Outcome: Percentage of Patients With Microbiological Improvement
Description: Percentage of patients with microbiological improvement, defined such that all bacteria present above threshold at Day 1 (Baseline) are eradicated (absent) or reduced at Day 7 based on a Classification of Microbial Response (Eradication=pathogen is absent in follow-up culture; Reduction=pathogen is reduced from baseline below threshold count in follow-up culture; Persistence=pathogen reduced from baseline but is above or equal to threshold count in follow-up culture; and Proliferation=pathogen has increased in count from baseline in follow-up culture).
Time Frame: Day 7
Population: as for outcome 1
Measure: Number; unit: Percentage of Patients
Arm/Group | Gatifloxacin 0.3% | Moxifloxacin 0.5%
Number analyzed (Participants) | 56 | 64
Percentage of Patients | 94.6 | 92.2

3. Secondary Outcome: Percentage of Patients With Improvement in Ocular Signs for Lid Erythema
Description: Percentage of patients with at least a 1-grade improvement in ocular signs for lid erythema at Day 7 from Day 1 (Baseline). Lid erythema was assessed on a 4-point severity grade scale (0=none, +1=mild, +2=moderate, +3=severe).
Time Frame: Days 7
Population: as for outcome 1
Measure: Number; unit: Percentage of Patients
Arm/Group | Gatifloxacin 0.3% | Moxifloxacin 0.5%
Number analyzed (Participants) | 56 | 64
Percentage of Patients | 76.8 | 75.0

4. Secondary Outcome: Percentage of Patients With Improvement in Ocular Signs for Conjunctival Discharge at Day 7
Description: Percentage of patients with at least a 1-grade improvement in ocular signs for conjunctival discharge at Day 7 from Day 1 (Baseline). Conjunctival discharge was assessed on a 4-point severity grade scale (0=none, +1=mild, +2=moderate,
  +3=severe).
Time Frame: Day 7
Population: as for outcome 1
Measure: Number; unit: Percentage of Patients
Arm/Group | Gatifloxacin 0.3% | Moxifloxacin 0.5%
Number analyzed (Participants) | 56 | 64
Percentage of Patients | 94.6 | 92.2

ADVERSE EVENTS:
Description: Safety Population used for SAE/AE analysis - defined as all patients who were randomized AND treated. Intent-to-Treat Population used for Participant Flow - defined as all patients who were randomized.
Arm/Group | Gatifloxacin 0.3% | Moxifloxacin 0.5%
Serious Adverse Events (participants affected / at risk) | 0/84 | 1/86
Other Adverse Events (participants affected / at risk) | 11/84 | 8/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gatifloxacin 0.3% (N=84) | Moxifloxacin 0.5% (N=86)
Pyrexia (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Gatifloxacin 0.3% (N=84) | Moxifloxacin 0.5% (N=86)
Conjunctivitis (Eye disorders) | 4 | 3
Conjunctivitis bacterial (Infections and infestations) | 7 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.